CLINICAL TRIAL: NCT06225960
Title: Dorsal Root Ganglion Stimulation: Assessment of Analgesic Efficacy in Postherpetic Neuropathy Based on Pain Phenotype
Brief Title: Dorsal Root Ganglion Stimulation in Postherpetic Neuropathy
Acronym: DRGs
Status: Enrolling by invitation | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Monaldi Hospital (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Nuovo Regina Margherita Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2360CE
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Postherpetic Neuralgia
Keywords: Postherpetic neuralgia, Dorsal root ganglion stimulation,
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is a prospective, multicenter observational study evaluating the efficacy of ganglion stimulation (medical device) in cases of post-herpetic neuropathy.

This study introduces recent methods of phenotypic stratification of postherpetic neuropathy into the field of interventional pain therapy. The aim is to identify which clinical expression of this diverse pathology can derive the greatest benefits from an otherwise effective but expensive therapy such as ganglion stimulation.

The study protocol includes the application of a common clinical practice, already in use for several years at the promoting center and participating centers (as well as internationally scientifically codified). It is supported by an innovative stratification of clinical expression (phenotype of the disease), recently introduced in the literature.

The study aims to identify, through careful clinical evaluation, predictive indices of the greatest success in invasive ganglion stimulation therapy, a treatment associated with significant system costs and considerable inconvenience for the patient.

The results of the experimentation will allow the codification of evaluative clinical pathways to predict a higher success index in certain clinical expressions of postherpetic neuropathy compared to others. This will help reduce the costs of implant trials and enable defining the real objective of the proposed therapy in consultation with the patient.

DETAILED DESCRIPTION:
During the manifestation of varicella, the varicella-zoster virus (VZV) localizes in the ganglia of dorsal roots or cranial nerves and remains latent until it can reactivate in conditions of reduced immunity, such as old age or certain diseases. Infection control is linked to cell-mediated immunity, which tends to decrease with age but can be periodically stimulated by exposure to chickenpox or silent reactivations..

Epidemiological studies demonstrate that herpes zoster affects 5.23 cases per 1000 persons/year, with 13.7% showing signs of postherpetic neuralgia (PHN) after three months. In individuals over 80 years, the PHN percentage rises to 80%. PHN is a very challenging-to-treat painful syndrome with diverse manifestations in patients.

During reactivation, the virus travels along the central and peripheral dendrites of the first neuron, reaching the skin where it causes vesicles, usually affecting a dermatome but sometimes more than one. Post-mortem histological studies have shown atrophy of the dorsal horns of the spinal cord and loss of cells, axons, and myelin in the dorsal root ganglion (DRG) of patients with long-lasting PHN; histopathological changes were confined to a single ganglion per patient. The loss of axons and myelin in sensory roots and nerves was also present in patients without pain. In some patients, a prolonged cell-mediated inflammatory process was evident .

Skin biopsy in PHN patients demonstrated a significant reduction in terminals of small-caliber fibers, more evident in the epidermis than in the dermis. The innervation of affected areas shows great variability among patients and is not correlated with pain intensity or the degree of allodynia.

At the molecular level, increased expression of voltage-sensitive Na+ channels, alterations in K+ channels, and an increase in transient receptor potential vanilloid 1 (TRPV1) have been demonstrated. These modifications alter the threshold for the generation of action potentials at the nerve terminals and can generate action potentials at the site of injury along the fiber or at the level of the DRG. There is also a postulated loss of inhibitory GABAergic interneurons in the dorsal horns and descending inhibition.

In a study investigating the correlation between neurophysiological tests and symptoms in patients with ophthalmic postherpetic neuralgia (PHN), Truini and colleagues demonstrated that the reduction in laser-evoked potentials (LEP) amplitude, due to the decrease in Aδ and C fibers, correlated with the intensity of continuous pain. On the other hand, abnormalities in the blink reflex, which assesses Aβ fibers, correlated with paroxysmal pain. Neurophysiological alterations did not correlate with the presence of allodynia.

Clinically, patients may experience spontaneous pain, predominantly burning, deep and dull, paroxysmal pain, and allodynia to mechanical and/or thermal stimuli. Some patients report unbearable itching (9). The various manifestations of signs and symptoms in patients with PHN suggest a spectrum of mechanisms:

1. Peripheral sensitization due to "irritable nociceptors," clinically characterized by spontaneous and evoked pain (allodynia) and few negative signs on evaluation; b) Partial loss of myelin and/or nerve fibers with spontaneous pain, allodynia, and areas of sensory deficit; c) Deafferentation with spontaneous pain, severe sensory deficits without allodynia.

   In all cases, there is sensitization of second-order neurons due to an excess of afferent impulses, modification of the connectivity of Aβ fibers, or loss of afferent impulses (deafferentation). In cases of extensive areas of sensory deficit, there may be a correspondence with histological pictures of widespread atrophy of dorsal horns, which also involve the somas of second-order neurons with deafferentation of the third-order neuron.

   Treatment of Postherpetic Neuralgia (PHN) The therapy for PHN involves topical and/or systemic pharmacological approaches with limited satisfaction, despite recent attempts to target therapies based on phenotypic considerations. Since pain is often poorly controlled by pharmacological treatment, various interventional neuromodulation techniques have been proposed for PHN treatment, ranging from more peripheral approaches (anesthetic and corticosteroid blocks on the peripheral nerve or paravertebral, radiofrequency modulation techniques, or cryoanalgesia) to those involving the ganglion (anesthetic and corticosteroid injection, pulsed radiofrequency modulation, radiofrequency lesion) or at the spinal cord level (spinal cord neurostimulation, spinal administration of drugs). The literature often reports clinical cases or case series.

   Given the frequent localization of PHN pain at the trunk level, the difficulty in achieving optimal paresthesia coverage of the pain area, and the involvement of a limited territory to one or a few nerve roots, dorsal root ganglion (DRG) stimulation has appeared as an interesting option in treating cases less responsive to pharmacological therapies and less invasive pain management techniques. In a poster presented at the first European INS congress, Pajuelo et al. reported a case series of 22 patients treated with DRG stimulation for PHN with encouraging results..

   Considering the diverse clinical presentations of PHN and the underlying pathogenetic mechanisms, it remains to be clarified which types of PHN patients are more likely to benefit from DRG stimulation and how to identify the ganglion(s) to be treated with neurostimulation.
   * the selected patients, subsequent to a clinical evaluation confirming the postherpetic origin of the painful condition, non-response to topical and systemic medications, and after defining the dermatomal area of neuropathy, the option of undergoing ganglion neurostimulation implantation will be proposed. This involves a preliminary trial phase with the potential for definitive implantation, similar to common clinical practice outside experimental protocols.

   The trial phase involves the implantation of a ganglion electrode (or electrodes in the case of multiple dermatomes) connected to an extracutaneous extension and linked to an external pulse generator (EPG). During the trial phase, the patient's clinical progress and response will be evaluated.

   At the conclusion of the trial phase, in the event of a positive response from the patient, definitive implantation will proceed through the placement of an internal pulse generator (IPG) via subcutaneous surgery at a location chosen by the operator. The decision for definitive implantation will be made in consultation with the patient, following common clinical practice, without specifying precise evaluation parameters to avoid limiting implantation opportunities for patients deciding to participate in the protocol compared to those normally treated (right to equitable care).

   T0 - Enrollment visit

   After the patient signs the consent form, the following tests will be administered:

   • Average minimum and maximum pain of the last month using the NRS scale (0-10) International scale to evaluate pain intensity
   * DN4 (Neuropatic Pain 4) in the validated Italian version;The items of the DN4 are scored based on a yes (1 point) /no (0 points) answer. This leads to a score range of 0-10 when the symptoms (range 0-7 points) as well as the signs (range 0-3 points) items are included.
   * SF12 (short form health questionnaire) in the validated Italian version; The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure
   * EQ5 (Euro QOL 5) in the validated Italian version. EQ-5D is an instrument which evaluates the generic quality of life developed in Europe

   In clinical examination, in accordance with the latest guidelines (14) for stratification through the evaluation of the sensory profile of patients with neuropathic pain, three categories (clusters) of patients will be identified:
   * "sensory loss": a signal of loss of small and large fibers, previously defined as deafferentation or hypoesthesia symptoms.
   * "thermal hyperalgesia": a sign of predominantly preserved large-diameter fibers and hyperalgesic response to heat and cold (previously described as "irritated nociceptor").
   * "mechanical hyperalgesia": loss of sensitivity to heat and cold due to small fiber deficits associated with pressure and pinprick hyperalgesia.

   At the end of this initial phase, depending on the enrolling center's clinical practice, the patient will be offered either an anesthetic block or pulsed ganglion neuromodulation to assess the patient's response. In the case of a clinically positive response, indicating short-term pain reduction or patient satisfaction (positive test but ineffective therapy), patients will be offered ganglion electrode implantation.

   T1: Ganglion electrode implantation (trial phase) During the trial phase, if the patient's dermatomal area has not been previously mapped using block and radiofrequency techniques, the level or levels of correspondence during sensory stimulation and the placement of the ganglion electrode will be evaluated. The definitive placement will be one where the electrode or electrodes are capable of generating "paresthesia" throughout the patient's painful area. In case it is not possible to achieve complete coverage (noting the reasons for such lack and estimating the percentage coverage), the ganglion electrode will be placed in the best possible position. If it is necessary to position the electrode catheters above and below the metamere (so-called "belting"), the patient will be considered a drop-out.

   T2: Evaluation of the trial phase at 1 month • Average minimum and maximum pain of the last month using the NRS scale (0-10);

   • DN4 (neuropathic pain) in the validated Italian version;

   • SF12 (short form health questionnaire) in the validated Italian version;

   • EQ5 (Euro QOL 5) in the validated Italian version;

   • PGIC (Patient Global Impression Change) with 7 items. T3: Clinical evaluation at 6 months (primary endpoint)

   At 6 months, patients who underwent definitive implantation will be administered the following tests by the physicians participating in the study:

   • Average minimum and maximum pain of the last month using the NRS scale (0-10);
   * DN4 (neuropathic pain) in the validated Italian version;
   * SF12 (short form health questionnaire) in the validated Italian version;
   * EQ5 (Euro QOL 5) in the validated Italian version;
   * PGIC (Patient Global Impression Change) with 7 items. .

   T4: Clinical evaluation at 12 months:

   At 12 months, patients who underwent definitive implantation will be administered the following tests by the physicians participating in the study:
   * Average minimum and maximum pain of the last month using the NRS scale (0-10);
   * DN4 (neuropathic pain) in the validated Italian version;
   * SF12 (short form health questionnaire) in the validated Italian version;
   * EQ5 (Euro QOL 5) in the validated Italian version;
   * PGIC (Patient Global Impression Change) with 7 items. The patient will also be reassessed by the physician who performed the initial evaluation to determine changes in response to the objective examination (pin-prick test, heat, cold, touch). In case of system removal between the 6th and 12th month, the reasons for removal (loss of efficacy, intolerance, etc.) will be recorded.

ELIGIBILITY:
Inclusion Criteria:•

* Subjects of both genders aged between 18 and 75 years;
* Patients with postherpetic neuralgia (PHN) for at least 6 months who have tried the topical and systemic pharmacological therapies recommended in the neuropathic pain guidelines
* Distribution of neuropathic pain in a region between C6 and L5;
* Individuals capable of adequately adhering to the study protocol and responding to the administered questionnaires;
* Signed informed consent.

Exclusion Criteria:

* Subjects with a history of major depression or other psychiatric conditions that, in the investigator's opinion, may interfere with study participation;
* Patients in presumed/confirmed pregnancy;
* Patients for whom the placement of spinal/ganglion stimulation systems is contraindicated due to systemic pathological conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with postherpetic neuralgia (PHN) for at least 6 months who have tried the topical and systemic pharmacological therapies recommended in the neuropathic pain guidelines
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-02-19 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Analgesic efficacy identifying the pathogenetic cluster with the greatest therapeutic response | at 6 months
  Average minimum and maximum pain with the NRS scale (0-10) DN4 (neuropathic pain) in the validated Italian version; SF12 (short form health questionnaire) in the validated Italian version• EQ5 (Euro QOL 5) in the validated Italian version.

CONTACTS AND LOCATIONS:
Locations (1):
- ICSMaugeri Spa, Pavia, Italy